CLINICAL TRIAL: NCT03546790
Title: Laboratory Smoking of Marijuana "Blunts"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Battelle Memorial Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BMI-104112
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Cannabis
Keywords: Cannabis
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Flavor 1 (Experimental): Grape flavored tobacco cigar wrapper
  Interventions: Drug: Marijuana
- Flavor 2 (Experimental): Chocolate flavored tobacco cigar wrapper
  Interventions: Drug: Marijuana
- Flavor 3 (Experimental): Tobacco flavored tobacco cigar wrapper
  Interventions: Drug: Marijuana

INTERVENTIONS:
Drug: Marijuana — Marijuana smoked via blunts with different cigar wrappers

SUMMARY:
This is a double-blind within-subjects clinical laboratory study comparing the product appeal and abuse liability-related subjective effects of different flavored cigar wrappers for marijuana blunts.

ELIGIBILITY:
Inclusion Criteria:

* Currently living in Baltimore City or Baltimore County, MD;
* Able to read, understand, and sign informed consent;
* 18-55 years old;
* Currently smokes marijuana blunts;
* Designation of Medically Healthy for Research by the Study Physician; and
* Willing to abstain from illicit drug use other than marijuana for the duration of the study.

Exclusion Criteria:

* BAC > 0.020% as measured by alcohol breathalyzer;
* Meets DSM-5 criteria for severe current or lifetime Cannabis Use Disorder;
* Meets DSM-5 criteria for any current Axis I disorder, other than current mild or moderate Cannabis Use Disorder;
* Self-reported current desire to stop marijuana use;
* Self-reported current asthma, chronic obstructive pulmonary disease, hypertension, cardiovascular disease or any other medical illness that precludes participation;
* Has difficulties with blood draws or poor venous access;
* History of blood donation in the past 30 days or receiving blood products within the past 2 months prior to any experimental visit;
* Among females, current pregnancy or lactation or attempting to get pregnant, or at risk of becoming pregnant;
* Acute illness which will require participant to be rescheduled

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Puff topography | During marijuana blunt smoking
  Total inhalation volume

SECONDARY OUTCOMES:
Carbon monoxide | Immediately after marijuana blunt smoking
  Exhaled breath carbon monoxide (ppm)
Subjective drug effects | Immediately after marijuana blunt smoking
  Ratings of "good" and "high"
Measures of demand | Immediately after marijuana blunt smoking
  Number of units an individual would purchase at varying price points

CONTACTS AND LOCATIONS:
Overall Officials: Wallace B Pickworth, PhD, Principal Investigator — Battelle Memorial Institute
Locations (1):
- Battelle Memorial Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No